CLINICAL TRIAL: NCT06227247
Title: Meals 4 Moms: Development and Feasibility of a Multilevel Community-based Lifestyle Intervention for Gestational Diabetes
Brief Title: Meals 4 Moms: A Multilevel Community-based Lifestyle Intervention for GDM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment pace was not sufficient to support fully-powered efficacy trial. Study investigators decided to terminate the feasibility trial before reaching recruitment target.
Sponsor: UConn Health (Other)
Collaborators: University of Connecticut (Other); Trinity Health Of New England (Other); Hartford Hospital (Other)
Responsible Party: Principal Investigator, Andrea Shields, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-190SSF-2
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes
Keywords: Diabetes; Gestational diabetes; Pregnancy; Exercise; Nutrition; Diabetes education
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: We plan to randomize 40 participants 1:1 to the M4M intervention vs usual GDM care (UC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meals 4 Moms intervention (Experimental): Participants randomized to the M4M condition will receive:
  * Food budget of $266 per week in credits to spend towards medically-tailored GDM meals
  * Enhanced educational GDM-specific education on exercise, nutrition, and blood sugar glucose management
  * Activity tracker and digital scale
  * Usual GDM care
  Interventions: Behavioral: Meals4Moms Intervention
- Usual GDM Care (No Intervention): Usual care (UC) will consist of the current treatment care that is provided by the participant's prenatal care provider. Usual care consists of a special diet, monitoring of blood glucose levels and encouragement/guidance of increasing a participant's exercise.

INTERVENTIONS:
Behavioral: Meals4Moms Intervention — A community-based, healthy living program including continued gestational diabetes (GDM) education, physical activity level monitoring, and delivery of medically-tailored GDM meals for the management of gestational diabetes in pregnant people.
  Arms: Meals 4 Moms intervention

SUMMARY:
The goal of the project is to conduct a pilot feasibility randomized trial comparing a community-based lifestyle intervention called Meals for Moms (M4M) versus the usual care for pregnant persons diagnosed with gestational diabetes (GDM). Participants will be randomly placed into the usual care (UC) comparison group or the M4M healthy living program, which includes continued GDM education, physical activity level monitoring, and delivery of medically-tailored GDM meals. The trial will assess if M4M is feasible for the management of gestational diabetes in pregnant patients.

DETAILED DESCRIPTION:
Gestational diabetes mellitus, or GDM, affects many pregnancies throughout the United States contributing to an increased risk of negative pregnancy outcomes such as delivery complications, hospitalizations, and poor clinical outcomes for both patients and infants. Additionally, many pregnant patients with GDM will progress to developing Type 2 diabetes within their lifetime. GDM, therefore, is the perfect window of opportunity for the prevention of diabetes.

GDM management requires education and adoption of a specific diet, daily blood sugar monitoring, exercise, and compliance with prenatal visits. Adopting all these changes may be hard to understand and comply with in a short window of time as, on average, patients are diagnosed GDM 8 to 10 before delivery. Thus, to achieve these goals quickly, patients must have immediate access to nutrient-rich food, and on-going education and support regarding healthy-meal preparation, including portion sizes, frequency, and composition of healthy snacking.

Previous and on-going research on health food prescription programs and supervised exercise sessions are often not performed with patients with GDM. To address this gap, investigators aim to develop a lifestyle intervention that promotes self-efficacy with unsupervised exercise and evidence-based behavioral strategies (e.g. goal setting, monitoring and feedback) and incorporate the use of physical activity tracking devices to support these strategies. This project has two distinct phases. First, to develop the novel Meals for Moms (M4M) community-based lifestyle intervention using feedback and input from women living with GDM. Second, to conduct a pilot feasibility randomized trial comparing the feasibility, compliance, and acceptability of the M4M intervention versus the usual care for pregnant persons diagnosed with GDM.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years old
* Current singleton pregnancy
* GDM diagnosis between 24+0 and 31+6 weeks gestation, and no more than 4weeks from time of diagnosis at time of enrollment.
* Currently receiving gestational diabetes management at the UConn Health Maternal Fetal Clinic, St. Francis's Hospital Women's Health clinic, Hartford Healthcare Women's Ambulatory Health Services (WAHS)
* Intends to deliver at either UConn Health, St. Francis Hospital or Hartford Healthcare
* Able to read and understand English well enough to participate in the study in English
* Daily access to the internet from smartphone, tablet computer, or laptop/desktop computer that they can use to participate in the study
* Medical clearance to participate from prenatal care provider including clearance to engage in physical activity
* Able to provide verbal or written consent for each component of the study procedures and data collection
* Currently lives within one of the meal delivery areas in Connecticut to allow for meal delivery (total of 32 eligible towns/cities)

Exclusion Criteria:

* Unable or unwilling to give informed consent or communicate with study staff.
* Diabetes mellitus (Type I or Type II).
* GDM diagnosed prior to 24 weeks gestation or after 32+0 weeks gestation.
* Patient is scheduled for a preterm delivery for medical reasons (i.e., placenta accreta, prior classical incision) at time of eligibility screening or at any time prior to randomization.
* Concurrent participation in another research study providing intervention related to GDM, pregnancy, diet, and/or physical activity.
* Medical conditions that may result in the inability to tolerate solid foods (i.e., hyperemesis gravidarum).
* Medical condition which would prohibit participation as indicated by prenatal care provider providing medical clearance.
* Dietary restrictions that cannot be accommodated for during meal preparation.
* Currently does not live in one of the towns listed within the meal delivery area.
* Has plans to move to out of the meal delivery area between enrollment and expected pregnancy due date.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Acceptability (participate again) | Follow-Up (within 2 weeks post-delivery)
  Percent of participants who report they would be likely or very likely to participate again if they had gestational diabetes (GDM) again.
Acceptability (recommended) | Follow-Up (within 2 weeks post-delivery)
  Percent of participants who report they would be likely to very likely to recommend the M4M intervention to a friend with gestational diabetes (GDM).
Recruitment | Baseline
  Recruitment rates will be calculated from the number of patients approached and reasons for ineligibility and non-participation.
Retention | Follow-Up (within 2 weeks post-delivery)
  Proportion of participants who complete any aspect of the follow-up assessment.
Receipt of intervention (Meal Ordering) | Follow-Up (within 2 weeks post-delivery)
  Percent of participants who spent at least 80% of weekly $260 food budget.
Receipt of intervention (Exercise Session Completion) | Follow-Up (within 2 weeks post-delivery)
  Percent of participants who completed at least 80% of exercise sessions they were eligible to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Shields, MD, MS, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Cosson E, Baz B, Gary F, Pharisien I, Nguyen MT, Sandre-Banon D, Jaber Y, Cussac-Pillegand C, Banu I, Carbillon L, Valensi P. Poor Reliability and Poor Adherence to Self-Monitoring of Blood Glucose Are Common in Women With Gestational Diabetes Mellitus and May Be Associated With Poor Pregnancy Outcomes. Diabetes Care. 2017 Sep;40(9):1181-1186. doi: 10.2337/dc17-0369. Epub 2017 Jul 19. PMID 28724718
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Berggren EK, Mele L, Landon MB, Spong CY, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Sciscione A, Catalano P, Harper M, Saade G, Caritis SN, Sorokin Y, Peaceman AM, Tolosa JE; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Perinatal outcomes in Hispanic and non-Hispanic white women with mild gestational diabetes. Obstet Gynecol. 2012 Nov;120(5):1099-104. doi: 10.1097/aog.0b013e31827049a5. PMID 23090528
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Chan CWH, Au Yeung E, Law BMH. Effectiveness of Physical Activity Interventions on Pregnancy-Related Outcomes among Pregnant Women: A Systematic Review. Int J Environ Res Public Health. 2019 May 23;16(10):1840. doi: 10.3390/ijerph16101840. PMID 31126153
- [Background] Garcia-Patterson A, Martin E, Ubeda J, Maria MA, de Leiva A, Corcoy R. Evaluation of light exercise in the treatment of gestational diabetes. Diabetes Care. 2001 Nov;24(11):2006-7. doi: 10.2337/diacare.24.11.2006. No abstract available. PMID 11679479
- [Background] Avery MD, Walker AJ. Acute effect of exercise on blood glucose and insulin levels in women with gestational diabetes. J Matern Fetal Med. 2001 Feb;10(1):52-8. doi: 10.1080/714904296. PMID 11332421
- [Background] Coe DP, Conger SA, Kendrick JM, Howard BC, Thompson DL, Bassett DR Jr, White JD. Postprandial walking reduces glucose levels in women with gestational diabetes mellitus. Appl Physiol Nutr Metab. 2018 May;43(5):531-534. doi: 10.1139/apnm-2017-0494. Epub 2017 Dec 22. PMID 29272606
- [Background] Onaade O, Maples JM, Rand B, Fortner KB, Zite NB, Ehrlich SF. Physical activity for blood glucose control in gestational diabetes mellitus: rationale and recommendations for translational behavioral interventions. Clin Diabetes Endocrinol. 2021 Apr 25;7(1):7. doi: 10.1186/s40842-021-00120-z. PMID 33896420
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Background] Hanson MA, Bardsley A, De-Regil LM, Moore SE, Oken E, Poston L, Ma RC, McAuliffe FM, Maleta K, Purandare CN, Yajnik CS, Rushwan H, Morris JL. The International Federation of Gynecology and Obstetrics (FIGO) recommendations on adolescent, preconception, and maternal nutrition: "Think Nutrition First". Int J Gynaecol Obstet. 2015 Oct;131 Suppl 4:S213-53. doi: 10.1016/S0020-7292(15)30034-5. No abstract available. PMID 26433230
- [Background] Chen TC, Clark J, Riddles MK, Mohadjer LK, Fakhouri THI. National Health and Nutrition Examination Survey, 2015-2018: Sample Design and Estimation Procedures. Vital Health Stat 2. 2020 Apr;(184):1-35. PMID 33663649
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Vandelanotte C, Spathonis KM, Eakin EG, Owen N. Website-delivered physical activity interventions a review of the literature. Am J Prev Med. 2007 Jul;33(1):54-64. doi: 10.1016/j.amepre.2007.02.041. PMID 17572313
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Hudson J, Nguku SM, Sleiman J, Karlen W, Dumont GA, Petersen CL, Warriner CB, Ansermino JM. Usability testing of a prototype Phone Oximeter with healthcare providers in high- and low-medical resource environments. Anaesthesia. 2012 Sep;67(9):957-67. doi: 10.1111/j.1365-2044.2012.07196.x. PMID 22861503
- [Background] Hordern MD, Dunstan DW, Prins JB, Baker MK, Singh MA, Coombes JS. Exercise prescription for patients with type 2 diabetes and pre-diabetes: a position statement from Exercise and Sport Science Australia. J Sci Med Sport. 2012 Jan;15(1):25-31. doi: 10.1016/j.jsams.2011.04.005. Epub 2011 May 28. PMID 21621458
- See also: A Subsidized Healthy Food Prescription Program for Adults With Type 2 Diabetes Who Are Experiencing Food Insecurity: Protocol for a Randomized Controlled Trial (PMCID: PMC8265448) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC8265448/